CLINICAL TRIAL: NCT01497015
Title: Memory Training Intervention for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Diane Von Ah, Associate Professor, Department Chair, School of Nursing, Indiana University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 64194
Record Dates: First submitted 2011-12-15; First posted 2011-12-22 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- memory training (Experimental): memory training 10 1-hour sessions with interventionist to be delivered over 6-8 weeks
  Interventions: Behavioral: memory training
- speed of processing training (Experimental): Speed of processing training 10 1-hour sessions delivered over 6-8 weeks
  Interventions: Behavioral: speed of processing training
- waitlist control (Experimental): Breast cancer survivors will be randomized to 1 of 3 groups: memory training, speed of process training or waitlist control
  Interventions: Behavioral: waitlist control

INTERVENTIONS:
Behavioral: memory training — 10 1-hour sessions over 6-8 weeks
  Arms: memory training
Behavioral: speed of processing training — 10 1-hour sessions delivered over 6-8 weeks
  Arms: speed of processing training
Behavioral: waitlist control — Breast cancer survivors will receive the speed of processing training compact disc in the mail after study completion.
  Arms: waitlist control

SUMMARY:
This is a randomized controlled trial to evaluate the ACTIVE memory training intervention and ACTIVE speed of processing training to waitlist, no-contact control conditions. Specific aims and hypotheses are:

Aim 1: Evaluate the acceptability and usefulness of the ACTIVE memory intervention among Breast Cancer Survivors (BCS).

Hypothesis 1: BCS assigned to the memory intervention arm will perceive the intervention as more acceptable and useful than BCS assigned to the attention control condition.

Aim 2: Establish preliminary efficacy of the ACTIVE memory training intervention relative to the attention control and no-contact control conditions.

Hypothesis 2: Memory training will result in greater memory enhancement immediately post and 2-months post-intervention relative to attention control or no-contact control conditions.

DETAILED DESCRIPTION:
Memory deficits are a prevalent, bothersome, and potentially debilitating symptom for millions of breast cancer survivors (BCS). Evidence-based treatment is difficult because there has been little intervention research in this area. Memory training may be a viable treatment option for BCS in need. Therefore, the purpose of this study is to examine the acceptability, usefulness, and preliminary efficacy of the memory training intervention from the Advanced Cognitive Training in Vital Elderly (ACTIVE) trial, the largest controlled trial of cognitive interventions in the behavioral sciences. The memory training intervention will be compared to attention control and no-contact control groups. Specific aims are to (1) evaluate the acceptability and usefulness of the memory intervention in BCS and (2) establish preliminary efficacy of the ACTIVE memory training intervention relative to attention control and no-contact control conditions. Acceptability and usefulness will be assessed through self-report. Memory will be assessed through objective neuropsychological tests. A total of 108 eligible BCS will be randomized to memory training, attention control, or no-contact control. A blinded and trained tester will perform data collection and neuropsychological testing at three time points: baseline prior to the intervention, immediately post-intervention, and 2 months post-intervention. Findings will provide information about the acceptability, usefulness, and preliminary efficacy of the ACTIVE memory training intervention on memory performance in BCS. Positive results will lead to a larger, full-scale study to determine efficacy of memory training interventions for BCS. Nursing interventional research in this area is vital to the development of evidence-based interventions to address memory deficits in BCS.

ELIGIBILITY:
Inclusion Criteria:

1. female gender (breast cancer is rare in men);
2. self-reported memory impairment and desire for treatment (to focus on BCS in greatest need);
3. first diagnosis of non-metastatic breast cancer (to control for multiple treatments or brain metastases in women with recurrent or metastatic disease);
4. ≥ 1 year post-treatment including surgery, radiation, and/or chemotherapy (reduce confounding factors related to acute effects of treatment);32
5. age ≥ 40 years (our prior studies indicate approximately 75% of BCS meet this criterion and reduce sample variability);
6. post-menopausal (majority are post-menopausal at diagnosis and reduce sample variability); and
7. able to read, write, understand, and speak English (to ensure informed consent).

Exclusion Criteria:

Women will be excluded if they have other co-morbidities or deficits that would sufficiently impair performance or inhibit cognitive training including:

1. substantial cognitive decline (score < 24 on the Mini Mental State Exam (MMSE);33
2. history of stroke, encephalitis, traumatic brain injury, brain surgery, dementia, Alzheimer disease, or Parkinson disease;
3. cranial radiation therapy or intrathecal therapy;
4. current active major depression or substance abuse or history of bipolar disorder, psychosis, schizophrenia, or learning disability;
5. history of or current other cancer except for basal cell skin cancer; or
6. receiving other cognitive training (to avoid exposure to other training).

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Memory Performance | Baseline, immediately post intervention
  Evaluate the acceptability and usefulness of the ACTIVE memory intervention among Breast Cancer Survivors.
Memory Performance | 2-month post intervention
  Evaluate the acceptability and usefulness of the ACTIVE memory intervention among Breast Cancer Survivors.

SECONDARY OUTCOMES:
Subjective Cognitive Function | baseline, immediately post intervention
  Preliminary efficacy established by objective neuropsychological tests and quality of life.
Subjective Cognitive Function | 2-month follow-up
  Post intervention efficacy established by objective neuropsychological tests and quality of life.
Symptom distress | baseline, immediately post intervention
  Preliminary symptom distress
Symptom distress | 2-month follow-up
  Post intervention symptom distress

CONTACTS AND LOCATIONS:
Overall Officials: Diane Von Ah, PhD, RN, CNA, Principal Investigator — Indiana University; Andrew Saykin, PsyD, Study Director — Indiana University; Frederick Unverzagt, PhD, Study Director — Indiana University; Janet Carpenter, PhD, RN, Study Director — Indiana University; Patrick Monahan, PhD, Study Director — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States